CLINICAL TRIAL: NCT00844155
Title: A Study of the Relative Oral Bioavailability of the Antiflu Medicine Oseltamivir (Tamiflu®) in Patients in the Intensive Care Unit
Brief Title: Study of the Relative Oral Bioavailability of the Antiflu Medicine Oseltamivir in the Intensive Care Unit
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study has been withdrawn as the H1N1 epidemic made this study redundant
Sponsor: University of Manitoba (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Principal Investigator, Dr. Faisal Siddiqui, Principal Investigator MD, University of Manitoba
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: #ML25018; Contract ID # 17908C
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Influenza A Virus Infection; Influenza B Virus Infection
Keywords: Prevention or treatment of influenza in ventilated patients
MeSH Terms: interventions — Oseltamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A.Oseltamivir 75 mg dose (Active Comparator): Patients will be randomized to two groups (group A) to receive oseltamivir at 75 mg, or (group B) to receive the drug at 150 mg in the fasting or fed state.
  Interventions: Drug: Oseltamivir 75 mg
- B. Oseltamivir 150mg (Active Comparator): Patients will be randomized to groups (group A) to receive oseltamivir at 75 mg, or group B to receive the drug at 150 mg in the fasting or fed state.
  Interventions: Drug: Oseltamivir 75 mg

INTERVENTIONS:
Drug: Oseltamivir 75 mg — The primary objective of this study is to demonstrate that the pharmacokinetics of oseltamivir, when given enterally to critically ill patients, in the standard treatment dose of 75 mg or double that dose, 150 mg, will yield a plasma concentration - versus - Time Area under the curve (AUC) similar to that observed in adults with influenza treated successfully with a dose of 75 mg, that the disposition characteristics are dose proportionate and are not altered by the concomitant administration of enteral feedings.
  Other Names: Tamiflu

SUMMARY:
This proposed pharmacokinetic study will test the hypothesis that in critically ill patients with respiratory failure requiring mechanical ventilation such as might be anticipated to be needed to treat patients with severe influenza pneumonia, oseltamivir administered enterally via nasogastric tube, with and without concomitant food or alimentation, will have similar oral bioavailability to that observed in ambulatory adults ill with influenza in whom oseltamivir therapy 75 mg BID is efficacious and well tolerated. Additionally, this experiment will test the hypothesis that increasing the dose (150 mg), with and without concomitant enteral feeding, will show a proportionate increase in bioavailability. Relative oral bioavailability will be assessed from plasma concentration vs. time over 12 hrs and urinary recovery of drug from 0 to 48 hrs after administration.

DETAILED DESCRIPTION:
Not required

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to the Intensive Care Unit requiring mechanical ventilation due to respiratory failure
* must be within the ages of 18-75 yrs

Exclusion Criteria:

* patients unable to have enteral feeding
* intolerance to oseltamivir
* pregnancy
* gastrointestinal or malabsorptive disease
* intestinal bypass surgery
* diarrhea (>2 loose bowel movements per day)
* receipt of prokinetic medications (metoclopramide, domperidone, erythromycin)
* severe liver disease (hepatocellular enzymes > 3 times the upper limit of normal)
* renal failure (Cockroft-Gault Creatinine Clearance < 30 ml/min, Dialysis dependant)
* cystic fibrosis
* intoxication or drug overdose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Oseltamivir administered enterally via nasogastric tube, with and without concomitant food or alimentation, will have similar oral bioavailability to that observed in ambulatory adults . | 13 months

SECONDARY OUTCOMES:
Test the hypothesis that increasing the dose (150 mg), with and without concomitant enteral feeding, will show a proportionate increase in bioavailability. | 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Faisal Siddiqui, MD, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada